CLINICAL TRIAL: NCT06842082
Title: A Multicenter, Prospective, Randomized, Single-blind Study Comparing Direct Laryngoscopy and Videolaryngoscopy for Orotracheal Intubation Performed by Anesthesia Residents in the Operating Room
Brief Title: The Videolaryngoscopy Versus Direct Laringoscopy for Residents Intubation Study
Acronym: VILARE-Adult
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario Lucus Augusti (Other)
Collaborators: Hospital Clinico Universitario de Santiago (Other); Complexo Hospitalario de Ourense (Other); Complejo Hospitalario Universitario de Pontevedra (Other); Complexo Hospitalario Universitario de A Coruña (Other); Complejo Hospitalario Universitario de Vigo (Other); Fundación de Investigación Biomédica - Hospital Universitario de La Princesa (Other); Hospital Arquitecto Marcide. Ferrol. A Coruña. (Spain) (Unknown)
Responsible Party: Principal Investigator, Maria Bermudez Lopez, Principal Investigator, Hospital Universitario Lucus Augusti
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: VILARE-Adults-Study
Record Dates: First submitted 2025-02-10; First posted 2025-02-24 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Intubation Intratracheal; Airway Management
Keywords: Intubation; anesthesia residents; videolaryngoscope; direct laryngoscope
MeSH Terms: interventions — Intubation

STUDY DESIGN:
Intervention Model Description: Laryngoscope Group: anesthesia resident intubation with Macintosh standard laryngoscope .
  Videolaryngoscope Group: anesthesia resident intubation with videolaryngoscope Mac-Style Blade.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laryngoscope Group (Active Comparator): For patients assigned to the Laryngoscope Group, the operator will use a Macintosh laryngoscope for the first laryngoscopy attempt
  Interventions: Device: Intubation with standard laryngoscope
- Videolaryngoscope Group (Active Comparator): For patients assigned to the Videolaryngoscope Group, the operator will use a videolaryngoscope with Mac-Style Blade for the first laryngoscopy attempt
  Interventions: Device: Intubation with video laryngoscope

INTERVENTIONS:
Device: Intubation with standard laryngoscope — Anesthesia resident will intubate using a standard laryngoscope.
  Arms: Laryngoscope Group
Device: Intubation with video laryngoscope — Anesthesia resident will intubate using a videolaryngoscope (Storz C-MAC, McGrath, Glidescope or other videolaryngoscope)
  Arms: Videolaryngoscope Group

SUMMARY:
The usual intubation technique in the operating room is based on direct laryngoscopy, using a standard Macintosh laryngoscope. However, this skill is not easy to acquire and requires adecuate training. Videolaryngoscopes are becoming a widely accepted airway management technique. because offer better view of the glottis and are easy to use. In addition, indirect laryngoscopes are useful for tracheal intubation by novice operators because of the feedback that supervisors can offer during intubation.

The goal of this clinical trial is to learn which intubation technique performed by residents of anesthesia in the operating room is better.

The main questions it aims to answer are:

* Which intubation technique is more effective for achieving first-attempt intubation?
* Which intubation technique results in fewer complications? Researchers will compare both intubation techniques performed by anesthesia residents in the operating room in adult anesthesia cases.

DETAILED DESCRIPTION:
The study will randomize, by means of a computer-generated randomization, approximately 1008 adults in two groups: Conventional group (Laryngoscope with Macintosh Blade) and Videolaryngoscope group (Mac-Style Blade) to be intubated in the operating room by an anesthesia resident.

Success rate of the selected technique (first attempt), overall success rate, number of attempts, complications, and duration of insertion for technique will be noted.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* Patients who need to be tracheal intubated for a surgical intervention in the surgical area.
* Intubation performed by an anesthesia resident.

Exclusion Criteria:

* Need for tracheal intubation with a device other than videolaryngoscopy or direct laryngoscopy (fiberoptic bronchoscope, tracheostomy...).
* Context of a Difficult Airway Management.
* Refusal of the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1008 (Estimated)
Dates: Start 2025-06-16 (Actual); Primary Completion 2025-12-29 (Estimated); Study Completion 2025-12-29 (Estimated)

PRIMARY OUTCOMES:
Difference in the first attempt success rate (percentage) | During intubation
  Success on the first attempt is defined as successfully passing the tube through the vocal cords in a single laryngoscopy attempt and inserting the endotracheal tube into the trachea

SECONDARY OUTCOMES:
Comparing the glottic view in the modified Cormack-Lehane scale between the two approaches | During intubation
  Modified Cormack-Lehane grade of glottic view:
  * I: full view of the glottis
  * IIa: partial view of the glottis
  * IIb: arytenoid or the posterior part of the vocal cords just visible
  * III: only epiglottis visible
  * IV: neither glottis nor epiglottis visible Cormack-Lehane grade of glottic view
Difference in percentage of "easy intubation" | During intubation
  To compare the difference in "easy intubation," defined as a Cormack-Lehane grade I-IIa glottic view and successful intubation on the first attempt, between the two intubation approaches.
Duration of laryngoscopy and tracheal intubation | During intubation
  The interval (in seconds) between the first insertion of a laryngoscope blade into the mouth and the final placement of a tube in the trachea.
Number of attempts to cannulate the trachea with an endotracheal tube | During intubation
  Number of attempts to cannulate the trachea with an endotracheal tube
Number of attempts to cannulate the trachea with a bougie. | During intubation
  Number of attempts to cannulate the trachea with a bougie
Need to change the device for intubation | During intubation
  Need to replace by another videolaryngoscope, a different angled blade, requirement for a fiberoptic bronchoscope...
Need for additional airway equipment | During intubation
  Airway equipment: bougie, stylet, other videolaryngoscope, others.
Operator-assessed difficulty of intubation | During intubation
  Operator-assessed difficulty of intubation
  * without difficulty
  * mild difficulty
  * moderate difficulty
  * severe difficulty
Use of external laryngeal pressure | During intubation
  External laryngeal pressure: Sellick maneuver or BURP
Reason for failure to intubate on the first attempt | During intubation
  Reason for failure among those who did not meet the primary outcome (successful intubation on the first attempt):
  * Inadequate view of the larynx
  * Inability to intubate the trachea with an endotracheal tube
  * Inability to cannulate the trachea with a bougie
  * Attempt aborted due to change in patient condition (e.g., worsening hypoxemia, hypotension, bradycardia, vomiting, bleeding)
  * Technical failure of the laryngoscope (e.g., battery, light source, camera, screen)
  * Other
Complications during intubation | Participants will be followed from the beginning of the intervention to 10 minutes after the intervention
  Complications during the procedure and within the following 10 minutes, including: hypotension (SBP < 80 mmHg), hypotension (SBP < 65 mmHg), O₂ saturation < 90%, O₂ saturation < 80%, bronchoaspiration, esophageal intubation, dental injury, airway injury, and others.

CONTACTS AND LOCATIONS:
Overall Officials: María Bermúdez María Bermúdez López, MD, Principal Investigator — Hospital Universitario Lucus Augusti
Locations (9):
- Spain (9):
  - Complejo Hospitalario Universitario de A Coruña, A Coruña, A Coruña
  - Hospital Universitario de Ferrol, Ferrol, A Coruña
  - Complejo Hospitalario Universitario de Santiago, Santiago, A Coruña
  - Hospital Universitario Lucus Agusti, Lugo, Lugo
  - Hospital Universitario de La Princesa, Madrid, Madrid
  - Complexo Hospitalario Universitario de Ourense, Ourense, Ourense
  - Complexo Hospitalario de Pontevedra, Pontevedra, Pontevedra
  - Complejo Hospitalario Alvaro Cunqueiro Vigo, Vigo, Pontevedra
  - Hospital POVISA de Vigo, Vigo, Pontevedra

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liu ZJ, Yi J, Guo WJ, Ma C, Huang YG. Comparison of McGrath Series 3 and Macintosh Laryngoscopes for Tracheal Intubation in Patients With Normal Airway by Inexperienced Anesthetists: A Randomized Study. Medicine (Baltimore). 2016 Jan;95(2):e2514. doi: 10.1097/MD.0000000000002514. PMID 26765472
- [Background] Taboada M, Estany-Gestal A, Rial M, Carinena A, Martinez A, Selas S, Eiras M, Veiras S, Ferreiroa E, Cardalda B, Lopez C, Calvo A, Fernandez J, Alvarez J, Alcantara JM, Seoane-Pillado T. Impact of Universal Use of the McGrath Videolaryngoscope as a Device for All Intubations in the Cardiac Operating Room. A Prospective Before-After VIDEOLAR-CAR Study. J Cardiothorac Vasc Anesth. 2024 Jul;38(7):1499-1505. doi: 10.1053/j.jvca.2024.03.016. Epub 2024 Mar 15. PMID 38580479
- [Background] Yamamoto Y, Kimura S, Kuniyoshi H, Hiroe T, Terui T, Kase Y. Novice residents' endotracheal intubation skill retention on a simulated mannequin after rotating at an anaesthesiology department: a randomized controlled study. J Int Med Res. 2023 Oct;51(10):3000605231206313. doi: 10.1177/03000605231206313. PMID 37848388
- [Derived] Taboada M, Bermudez M, Fernandez J, Estany-Gestal A, Jose Amate J, Ruido R, Amor M, Mato R, Barreiro C, Martinez P, Ramasco F, Vazquez O, Seoane-Pillado T. Videolaryngoscopy versus Direct Laryngoscopy for Tracheal Intubation by Anesthesia Residents in the operating room: the Randomized Multicenter VILARE Trial Protocol. Rev Esp Anestesiol Reanim (Engl Ed). 2026 Jan 12:501988. doi: 10.1016/j.redare.2026.501988. Online ahead of print. PMID 41534770